CLINICAL TRIAL: NCT05797103
Title: A Novel Electrolyzed Water Spray Reduces the Number of Bacteria E-coli and an Attenuated Human Flu Virus on Human Hands
Brief Title: The Research of Novel Electrolyzed Water Spray to Eradicate Bacteria E-coli and an Attenuated Human Flu Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jia19961018
Record Dates: First submitted 2023-02-27; First posted 2023-04-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Growth; Novel Influenza A (H1N1)
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; E-coli; Human flu virus
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Masking Description: This is an open label, two arm clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electrolyzed water spray group (Experimental): Participants with bacteria E-coli and an attenuated human flu virus on their hands will receive one treatment with the novel electrolyzed water and complete the questionnaire.
  Interventions: Device: A novel electrolyzed water spray reduces numbers of bacteria E-coli and an attenuated human flu virus on human hands
- untreated tap water group (Experimental): Participants with bacteria E-coli and an attenuated human flu virus on their hands will receive one treatment with the untreated tap water and complete the questionnaire.
  Interventions: Device: A novel electrolyzed water spray reduces numbers of bacteria E-coli and an attenuated human flu virus on human hands

INTERVENTIONS:
Device: A novel electrolyzed water spray reduces numbers of bacteria E-coli and an attenuated human flu virus on human hands — Electrolyzed water spray group will use the novel electrolyzed water spray to flush the hands that daub E. coli and attenuated human influenza virus H1N1 for 6 seconds per hand, and then use 4 seconds to collect a sample of the water flowing from the sprayed hand and apply it to the plate. Untreated tap water group will use the untreated tap water spray to flush the hands that daub E. coli and attenuated human influenza virus H1N1 for 6 seconds per hand, and then use 4 seconds to collect a sample of the water flowing from the sprayed hand and apply it to the plate.

SUMMARY:
The purpose of this study is to test whether spraying the hand of patients by use of the novel electrolyzed water spray will decrease the number of bacteria E-coli and the virus titer of an attenuated human flu virus.

DETAILED DESCRIPTION:
In this study, water including tap water, pure water and salt water, and an apparatus for producing electrolyzed water were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential（ORP）≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of dissolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion. The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U).

In this study, we hypothesize that the instantly generated electrolyzed water mist spray or spray relieves skin and mucosal inflammation including the itches through indirect actions by killing microbials and reducing endotoxin level and direct action by serving as an inflammatory inhibitor.

Detection of residual E. coli in the collected water samples. 1 ml of the collected water sample is inoculated on the surface of the solid LB agar plates and cultured overnight at 37°C in an incubator. Calculate the total number of bacterial colonies as CFU. In other words, the total number of bacteria/ml inoculated water sample (CFU) is the number of colonies formed on the surface of the plate. It is assumed that the bacteria on the hands are mostly washed out into the drain water sample pool and that the left over bacteria on the hand after rinsing is negligible. The leftover also can be measured by pressing the rinsed hand after on a large LB agar plate and then count the colonies (unstained and stained) after overnight incubation at 37°C.

Detection of residual human influenza virus H1N1 titers in the collected water samples. Viral titer (TCID50) is used to measure the infection of the dosage of 50% MDCK cells. MDCK cells were inoculated into 96-well plates at 1.0×104 cells per well and cultured overnight at 37°C in a cell culture incubator. We wash the hands and collect the drained water for the titer measurement. 100 ul of the water sample after the multiple proportion dilutions is inoculated into 96-well plates which contain overnight cultured MDCK cells. After 3 days of incubation at 37°C, TCID50 was calculated using the Reed and Muench method. 1 plaque forming unit (PFU) is equal to 1 alive virus particle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Male or female of any race and ethnicity.
3. Subject agrees to comply with study requirements.

Exclusion Criteria:

1. Severely unhealthy participants.
2. 80 years or older.
3. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
4. Dermatologic disease such as psoriasis or atopic dermatitis which may have inherently abnormal antimicrobial peptide levels.
5. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier.
6. Immunocompromised subjects, or with a history of active or malignant disease as determined by the participant's medical history.
7. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
8. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Flush and eradicate the number of bacteria E-coli on human hands. | 10 seconds
  Calculate the total number of bacterial colonies formed, expressed as CFU, and the total number of bacterial colonies (CFU) is the total number of colonies formed on the surface of a solid medium in 1 ml of a water sample.
  Viral titer (TCID50) indicates the minimum number of bacteria or amount of toxin required to infect half of an animal of a certain body weight or age by a specified route of infection within a specified time.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: No